CLINICAL TRIAL: NCT02263872
Title: Minocycline as an Adjunct for the Treatment of Depressive Symptoms: Pilot Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MINDEP001
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Depressive Disorder; Mood Disorders; Depressive Disorder, Treatment Resistant; Antidepressive Agents
MeSH Terms: conditions — Depressive Disorder; Mood Disorders; Depressive Disorder, Treatment-Resistant | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental): Minocycline 200mg perday
  Interventions: Drug: Minocycline
- comparison group with placebo (Placebo Comparator): Placebo provide
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 200mg perday
  Other Names: mesodrum

SUMMARY:
In this double blind randomised controlled pilot trial the investigators aim to determine the efficacy of minocycline as an adjunct to treatment as usual in patients with major depressive disorder. The investigators hypothesize that the multiple neuroprotective effects of minocycline will lead to an improvement in depressive symptoms in participants that were given minocycline plus treatment as usual

DETAILED DESCRIPTION:
Major depressive disorder is associated with significant morbidity and mortality. According to the WHO, depression is the leading cause of disability worldwide in terms of years lost due to disability [1]. Although depressive symptoms are amenable to antidepressant treatment, a high proportion of patients does not respond or remit. For example in the Sequenced Treatment Alternatives for the Relief of Depression (STAR*D) study the response and remission rates with stage 1 treatment (citalopram) were 49% and 37% respectively and these rates decreased to 16% and 13% respectively over the subsequent next three treatment steps [2]. Clearly there is a need for new treatment approaches.

Recently there has been significant preclinical and clinical study linking inflammatory processes to a range of psychiatric illness including depression, schizophrenia, bipolar disorder and Alzheimer's disease. The evidence that depression is an inflammatory related disorder comes from multiple sources. Depression is associated with raised inflammatory markers even in the absence of a medical illness [3]. More specifically depression has been associated with higher levels of positive acute phase proteins (APPs) and low levels of negative APPs [4] as well as increased levels of complement factors C3c and C4 and immunoglobulin M (IgM) and IgG [5]. Inflammatory medical illness, both CNS and peripheral, are associated with greater rates of depression. In patients with Crohns disease and comorbid depression bouts of physical disease activity tend to co-occur with depressive episodes [6]. Finally, patients treated with cytokines for various illnesses have an increased risk of developing depressive illness [7]. For example, treatment with cytokine IFN-α leads to the development of depressive symptoms in up to 45% of patients [8].

With this in mind it would seem logical to hypothesise that the addition of an anti-inflammatory medication may be a treatment option in depressive illness. Muller et al [9] were successful in showing this when they used Celcoxib in addition to Reboxetine for the treatment of major depressive disorder in a double-blind, randomised, placebo-controlled pilot study. Other studies have shown that TNF (tumour necrosis factor) blocking agents such as Infliximab and Ethanercept improve mood independent of improvement in inflammatory condition [10]. However some studies have found that anti-inflammatories may in fact have an antagonistic effect on the antidepressant actions of SSRIs [11]. Further work is needed in this area to clarify the role of inflammatory processes and anti-inflammatories in the treatment of depression.

Alongside the current interest in the use of anti-inflammatories as novel treatments in psychiatric illness, the antibiotic minocycline has also been proposed for the treatment of depressive symptoms as well as negative symptoms in schizophrenia [12, 13]. Preliminary data from an open label study of patients with psychotic unipolar depression also suggested that minocycline augmentation of antidepressant treatment was effective and well tolerated [14]. Minocycline is a pleiotropic agent that exerts effects on multiple interacting symptoms (e.g. anti-inflammatory, anti-oxidant, anti-apoptotic, anti-gutamatergic, monaminergic) implicated in the pathophysiology of mood disorders. Despite such neuroprotective properties, there have been no clinical trials to date investigating the antidepressant effects of minocycline in individuals. The investigators have previously shown that the addition of minocycline to treatment as usual early in the course of schizophrenia leads to a predominant improvement in negative symptoms.

In this double blind randomised controlled pilot trial the investigators aim to determine the efficacy of minocycline as an adjunct to treatment as usual in patients with major depressive disorder. The investigators hypothesise that the multiple neuroprotective effects of minocycline will lead to an improvement in depressive symptoms in participants that were given minocycline plus treatment as usual.

Aim To investigate whether the addition of minocycline to treatment as usual (TAU) for 3 months in patients with major depressive disorder will lead to an improvement in depressive symptoms compared with TAU.

Methods

Double blind randomised, placebo-controlled pilot trial.

The study will be conducted in Karachi, Pakistan. Patients will be recruited from psychiatric units in Karachi. All patients will give written informed consent after reading information in Urdu, witnessed almost always by a relative.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 18-65 years
2. Diagnostic and Statistical Manual-IV (DSM-IV) diagnosis of major depressive disorder
3. competent and willing to give informed consent
4. taking the current antidepressant medication for a minimum of 4 weeks prior to baseline
5. the current episode of depression has failed to remit with at least two courses of antidepressant treatment (one of which is the current course)
6. able to take oral medication
7. if female, willing to use adequate contraceptive precautions and to have monthly pregnancy tests.

Exclusion Criteria:

1. relevant medical illness (renal, hepatic, cardiac, serious dermatological disorders such as exfoliative dermatitis, systemic lupus erythematosis)
2. prior history of intolerance to any of the tetracyclines
3. concomitant penicillin therapy
4. concomitant anticoagulant therapy
5. presence of a seizure disorder
6. currently taking valproic acid
7. any change of psychotropic medications within the previous 4 weeks
8. diagnosis of substance abuse (except nicotine or caffeine) or dependence within the last 3 months according to DSM-IV criteria
9. pregnant or breast-feeding
10. presence of primary psychotic disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The primary clinical outcome measures will be mean change from baseline on the Hamilton Depression Scale scores | 12 weeks

SECONDARY OUTCOMES:
PHQ-9 | Baseline, Week 2, week 4, week 8, week 12
GAD-7 | Baseline, Week 2, week 4, week 8, week 12
CGI | Baseline, Week 2, week 4, week 8, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Muhammad Ishrat, Principal Investigator — Institute of Psychiatry, Psychology and Neuroscience, Kings college London
Locations (3):
- Pakistan (3):
  - Abasi Shaheed Hospital, Karachi, Sindh
  - Civil hospital Karachi, Karachi, Sindh
  - Karwan-e-Hayat, Karachi, Sindh

REFERENCES:
- [Background] World Health Organization. The Global Burden of Disease. Geneva: WHO Press; 2012.
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] O'Donovan A, Rush G, Hoatam G, Hughes BM, McCrohan A, Kelleher C, O'Farrelly C, Malone KM. Suicidal ideation is associated with elevated inflammation in patients with major depressive disorder. Depress Anxiety. 2013 Apr;30(4):307-14. doi: 10.1002/da.22087. Epub 2013 Mar 15. PMID 23504697
- [Background] Dantzer R, O'Connor JC, Freund GG, Johnson RW, Kelley KW. From inflammation to sickness and depression: when the immune system subjugates the brain. Nat Rev Neurosci. 2008 Jan;9(1):46-56. doi: 10.1038/nrn2297. PMID 18073775
- [Background] Song C, Dinan T, Leonard BE. Changes in immunoglobulin, complement and acute phase protein levels in the depressed patients and normal controls. J Affect Disord. 1994 Apr;30(4):283-8. doi: 10.1016/0165-0327(94)90135-x. PMID 7516941
- [Background] Mardini HE, Kip KE, Wilson JW. Crohn's disease: a two-year prospective study of the association between psychological distress and disease activity. Dig Dis Sci. 2004 Mar;49(3):492-7. doi: 10.1023/b:ddas.0000020509.23162.cc. PMID 15139504
- [Background] Van Gool AR, Kruit WH, Engels FK, Stoter G, Bannink M, Eggermont AM. Neuropsychiatric side effects of interferon-alfa therapy. Pharm World Sci. 2003 Feb;25(1):11-20. doi: 10.1023/a:1022449613907. PMID 12661471
- [Background] Capuron L, Miller AH. Immune system to brain signaling: neuropsychopharmacological implications. Pharmacol Ther. 2011 May;130(2):226-38. doi: 10.1016/j.pharmthera.2011.01.014. Epub 2011 Feb 17. PMID 21334376
- [Background] Muller N, Schwarz MJ, Dehning S, Douhe A, Cerovecki A, Goldstein-Muller B, Spellmann I, Hetzel G, Maino K, Kleindienst N, Moller HJ, Arolt V, Riedel M. The cyclooxygenase-2 inhibitor celecoxib has therapeutic effects in major depression: results of a double-blind, randomized, placebo controlled, add-on pilot study to reboxetine. Mol Psychiatry. 2006 Jul;11(7):680-4. doi: 10.1038/sj.mp.4001805. Epub 2006 Feb 21. PMID 16491133
- [Background] Krishnadas R, Cavanagh J. Depression: an inflammatory illness? J Neurol Neurosurg Psychiatry. 2012 May;83(5):495-502. doi: 10.1136/jnnp-2011-301779. Epub 2012 Mar 15. PMID 22423117
- [Background] Warner-Schmidt JL, Vanover KE, Chen EY, Marshall JJ, Greengard P. Antidepressant effects of selective serotonin reuptake inhibitors (SSRIs) are attenuated by antiinflammatory drugs in mice and humans. Proc Natl Acad Sci U S A. 2011 May 31;108(22):9262-7. doi: 10.1073/pnas.1104836108. Epub 2011 Apr 25. PMID 21518864
- [Background] Soczynska JK, Mansur RB, Brietzke E, Swardfager W, Kennedy SH, Woldeyohannes HO, Powell AM, Manierka MS, McIntyre RS. Novel therapeutic targets in depression: minocycline as a candidate treatment. Behav Brain Res. 2012 Dec 1;235(2):302-17. doi: 10.1016/j.bbr.2012.07.026. Epub 2012 Aug 10. PMID 22963995
- [Background] Chaudhry IB, Hallak J, Husain N, Minhas F, Stirling J, Richardson P, Dursun S, Dunn G, Deakin B. Minocycline benefits negative symptoms in early schizophrenia: a randomised double-blind placebo-controlled clinical trial in patients on standard treatment. J Psychopharmacol. 2012 Sep;26(9):1185-93. doi: 10.1177/0269881112444941. Epub 2012 Apr 23. PMID 22526685
- [Background] Miyaoka T, Furuya M, Yasuda H, Hayashida M, Nishida A, Inagaki T, Horiguchi J. Yi-gan san as adjunctive therapy for treatment-resistant schizophrenia: an open-label study. Clin Neuropharmacol. 2009 Jan-Feb;32(1):6-9. doi: 10.1097/WNF.0b013e31817e08c3. PMID 19471183
- [Derived] Zazula R, Husain MI, Mohebbi M, Walker AJ, Chaudhry IB, Khoso AB, Ashton MM, Agustini B, Husain N, Deakin J, Young AH, Berk M, Kanchanatawan B, Ng CH, Maes M, Berk L, Singh AB, Malhi GS, Dean OM. Minocycline as adjunctive treatment for major depressive disorder: Pooled data from two randomized controlled trials. Aust N Z J Psychiatry. 2021 Aug;55(8):784-798. doi: 10.1177/0004867420965697. Epub 2020 Oct 22. PMID 33092404
- [Derived] Husain MI, Chaudhry IB, Husain N, Khoso AB, Rahman RR, Hamirani MM, Hodsoll J, Qurashi I, Deakin JF, Young AH. Minocycline as an adjunct for treatment-resistant depressive symptoms: A pilot randomised placebo-controlled trial. J Psychopharmacol. 2017 Sep;31(9):1166-1175. doi: 10.1177/0269881117724352. Epub 2017 Aug 31. PMID 28857658
- [Derived] Husain MI, Chaudhry IB, Rahman RR, Hamirani MM, Qurashi I, Khoso AB, Deakin JF, Husain N, Young AH. Minocycline as an adjunct for treatment-resistant depressive symptoms: study protocol for a pilot randomised controlled trial. Trials. 2015 Sep 15;16:410. doi: 10.1186/s13063-015-0933-5. PMID 26374703